CLINICAL TRIAL: NCT02368951
Title: An Open-label,Phase I, Dose-escalation Trial to Evaluate the Safety, Tolerability, Maximum Tolerated Dose, Pharmacokinetic, and Pharmacodynamics of the Anti-FGFR2 Antibody Drug Conjugate BAY1187982 in Subjects With Advanced Solid Tumors Known to Express FGFR2.
Brief Title: Phase I, Dose-escalation Trial of BAY1187982 in Subjects With Advanced Solid Tumors Known to Express Fibroblast Growth Factor Receptor 2 (FGFR2)
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 16897
Record Dates: First submitted 2015-02-16; First posted 2015-02-23 (Estimated); Last update posted 2017-07-12 (Actual); Status verified 2017-07

CONDITIONS: Medical Oncology
Keywords: Phase 1; Solid Tumors; FGFR2; Antibody drug conjugate
MeSH Terms: interventions — aprutumab ixadotin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- BAY1187982 (Experimental): Dose-escalation phase:
  Approximately 30 subjects will participate in the dose-escalation phase The total number of subjects will depend on the number of cohorts necessary to identify the MTD.
  MTD expansion phase:
  Once the MTD has been determined, two expansion cohorts in FGFR2 expressing indications are planned:
  Cohort 1: Triple negative breast cancer (TNBC). This cohort will enroll 80 subjects (N=40 with low to moderate FGFR2 expression and N=40 with high FGFR2 expression) Cohort 2: Other indications expressing FGFR2. This cohort 40 subjects will be enrolled.
  Interventions: Drug: BAY1187982

INTERVENTIONS:
Drug: BAY1187982 — A dose of 0.1 mg BAY 1187982 per kilogram (kg) body weight (BW) was chosen as the starting dose based on toxicology data. The investigational drug will be administered as a 1-hour IV infusion once every 21 days at the trial site (Day 1 of each 21-day Cycle). The maximum possible dose escalation will be 2-fold and not more than 0.5 mg/kg BW until maximum tolerated dose is selected

SUMMARY:
To evaluate the safety, tolerability, maximum tolerated dose, pharmacokinetics, and pharmacodynamics of the anti-FGFR2 antibody drug conjugate BAY1187982 in subjects with advanced solid tumors known to express fibroblast growth factor receptor 2 (FGFR2)

ELIGIBILITY:
Inclusion Criteria:

* All subjects must be >/= 18 years at the first screening examination / visit
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1
* Subjects with advanced, histologically or cytologically confirmed solid tumors described to express fibroblast growth factor receptor 2 (FGFR2) that are refractory to any standard therapy
* For maximum tolerated dose (MTD) Dose Expansion: Subjects with advanced, histologically or cytologically confirmed triple-negative breast cancer who had undergone within 4 lines of systemic anti-cancer treatment and not eligible for standard therapy anymore.
* Subjects need to have evaluable disease (measurable or not measurable).
* Women of childbearing potential must have a negative pregnancy test performed within 7 days prior to the start of treatment

Exclusion Criteria:

* History of allergic reactions to monoclonal antibody therapy (or excipients in the formulation)
* Anti-cancer chemotherapy, experimental cancer therapy including clinical trial, or cancer immunotherapy within 4 weeks prior to the first dose of the investigational drug.
* Toxic effects of previous anti-cancer chemotherapy, experimental cancer therapy, or cancer immunotherapy have not normalized.
* History of symptomatic metastatic brain or meningeal tumors unless the subject is longer than 3 months from the end of definitive therapy before the first dose of the investigational drug and has clinically or radiologically no evidence of tumor growth.
* History of clinically significant cardiac disease
* Congenital coagulation abnormalities
* Subjects who are pregnant or are breast-feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2015-03-24 (Actual); Primary Completion 2016-07-27 (Actual); Study Completion 2016-07-27 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose(MTD) | Up to 2 years
  The MTD is defined as the maximum dose at which the incidence of DLTs during Cycle 1 is below 20%, or the maximum dose administered, whichever is achieved first during dose escalation
Number of subjects with adverse events as a measure of safety and tolerability | Up to 2 years
Number of subjects with serious adverse events as a measure of safety and tolerability | Up to 2 years

SECONDARY OUTCOMES:
Cmax (maximum observed drug concentration in measured matrix after single dose administration) | Cycles 1 and 3, Day 1: pre-dose, end of infusion, Day 2, Day 3, Day 5, Day 8, and Day 15.Cycles 2 and 4: Day 1: pre-dose.Cycle 5 Day 1 and every odd cycles after: pre-dose and end of infusion
AUC(0-tlast) AUC from time 0 to the last data point >LLOQ | Cycles 1 and 3, Day 1: pre-dose, end of infusion, Day 2, Day 3, Day 5, Day 8, and Day 15.Cycles 2 and 4: Day 1: pre-dose.Cycle 5 Day 1 and every odd cycles after: pre-dose and end of infusion
AUC)0-504 (AUC from zero to 504 hours post infusion) | Cycles 1 and 3, Day 1: pre-dose, end of infusion, Day 2, Day 3, Day 5, Day 8, and Day 15.Cycles 2 and 4: Day 1: pre-dose.Cycle 5 Day 1 and every odd cycles after: pre-dose and end of infusion
AUC (area under the concentration vs. time curve from zero to infinity after single (first) | Cycles 1 and 3, Day 1: pre-dose, end of infusion, Day 2, Day 3, Day 5, Day 8, and Day 15.Cycles 2 and 4: Day 1: pre-dose.Cycle 5 Day 1 and every odd cycles after: pre-dose and end of infusion
Cmax,md (maximum observed drug concentration in measured matrix after multiple dose administration during a dosage interval) | Cycles 1 and 3, Day 1: pre-dose, end of infusion, Day 2, Day 3, Day 5, Day 8, and Day 15.Cycles 2 and 4: Day 1: pre-dose.Cycle 5 Day 1 and every odd cycles after: pre-dose and end of infusion
AUC(0-tlast)md (AUC from time 0 to the last data point >LLOQ after multiple dosing) | Cycles 1 and 3, Day 1: pre-dose, end of infusion, Day 2, Day 3, Day 5, Day 8, and Day 15.Cycles 2 and 4: Day 1: pre-dose.Cycle 5 Day 1 and every odd cycles after: pre-dose and end of infusion
AUC(0-504)md | Cycles 1 and 3, Day 1: pre-dose, end of infusion, Day 2, Day 3, Day 5, Day 8, and Day 15.Cycles 2 and 4: Day 1: pre-dose.Cycle 5 Day 1 and every odd cycles after: pre-dose and end of infusion
FGFR2 levels in tumor tissue sample | Screening
CK18 levels in tumor tissue sample | Screening, Cycles 1 and 3, Day 1: pre-dose, end of infusion, Day 2, Day 3, Day 5, Day 8, and Day 15.Cycles 2 and 4: Day 1: pre-dose and end of infusion.
Nucleosome level in plasma | Screening, Cycles 1 and 3, Day 1: pre-dose, end of infusion, Day 2, Day 3, Day 5, Day 8, and Day 15.Cycles 2 and 4: Day 1: pre-dose and end of infusion.
Development of anti-drug antibodies (ADAs) in plasma as an indicator of immunogenicity | Cycle 1: Day 1: before infusion (pre-dose), Day 8
Tumor response | Screening, Day 15 (± 7 days) of Cycle 2 and every even subsequent Cycle (i.e. Cycles 2, 4, 6, 8, etc.)

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (12):
- United States (10):
  - San Francisco, California
  - Santa Monica, California
  - New Haven, Connecticut
  - Chicago, Illinois
  - Baltimore, Maryland
  - St Louis, Missouri
  - New York, New York
  - Nashville, Tennessee
  - Houston, Texas
  - Seattle, Washington
- Singapore, Singapore
- Seoul, South Korea

REFERENCES:
- [Derived] Kim SB, Meric-Bernstam F, Kalyan A, Babich A, Liu R, Tanigawa T, Sommer A, Osada M, Reetz F, Laurent D, Wittemer-Rump S, Berlin J. First-in-Human Phase I Study of Aprutumab Ixadotin, a Fibroblast Growth Factor Receptor 2 Antibody-Drug Conjugate (BAY 1187982) in Patients with Advanced Cancer. Target Oncol. 2019 Oct;14(5):591-601. doi: 10.1007/s11523-019-00670-4. PMID 31502117